CLINICAL TRIAL: NCT01298609
Title: A Randomized Controlled Pilot Study to Examine the Efficacy of Greater Occipital Nerve (C2) Stimulation in the Treatment of Fibromyalgia
Brief Title: Occipital Nerve (C2) Stimulation in the Treatment of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRD_545
Record Dates: First submitted 2011-02-14; First posted 2011-02-17 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Occipital Nerve Stimulation
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Suprathreshold Stimulation (Active Comparator): Patients will be stimulated at supra-sensory threshold levels for two weeks using occipital stimulation
  Interventions: Device: Occipital Stimulation
- minimal stimulation (Sham Comparator): Patients will be stimulated at minimal stimulation for two weeks using occipital stimulation
  Interventions: Device: Occipital Stimulation
- Subthreshold Stimulation (Active Comparator): Patients will be stimulated at sub-sensory threshold stimulation for two weeks using occipital stimulation
  Interventions: Device: Occipital Stimulation

INTERVENTIONS:
Device: Occipital Stimulation — Occipital Nerve Stimulation will be used in each study arm using the Eon Mini neuromodulation system

SUMMARY:
The study is designed as a prospective, randomized, double-blind, single center study with a 6 month duration post permanent system implantation. Forty patients will be implanted.

During trial stimulation, patients will be randomized into one of two study arms for two weeks. Crossover will occur at the 2 week study visit to the opposite group. After completion of these two arms, every patient will subsequently complete participation in the third study arm.

After completion of the third arm, patients will be evaluated to determine if they are a positive responder responder. If so, the patient will have the option of obtaining the permanent implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to provide informed consent to participate in the study;
2. Patient has had chronic widespread pain for at least 3 months in all 4 body quadrants;
3. Patient has at least 11 out of 18 tender points based on the tender points examination;
4. Patient has attempted "best" medical therapy and has tried and failed at least three documented medically supervised treatments (including, but not limited to drugs, physical therapy, acupuncture, etc.);
5. Patient medication has remained stable for at least 4 weeks prior to baseline data collection;
6. Psychological screening has been completed and the patient has been cleared by a psychologist as a suitable study candidate;
7. Patient agrees not to add or increase medication throughout the randomization trial period of the study;
8. Patient is willing to cooperate with the study requirements including compliance with the treatment regimen and completion of all office visits.

Exclusion Criteria:

1. Patient has current evidence of any psychiatric disorder, as documented by the DSM-IV-TR criteria with psychotic characteristics, (e.g. bipolar disorder, major depressive disorder);
2. Patient has been diagnosed with any disease mimicking the symptoms of the Fibromyalgia Syndrome (e.g. Epstein Barr, autoimmune diseases, etc.) that is not currently being treated or has not been stable for at least 6 months;
3. Patient is currently in active menopause;
4. Patient has been diagnosed with sleep apnea and is not currently involved in a treatment regime;
5. Patient has a history of substance abuse or substance dependency in the past 6 months prior to baseline data collection;
6. Patient currently participating in another clinical study;
7. Patient with demand-type cardiac pacemakers, an infusion pump or any implantable neurostimulator device;
8. Patient is likely to require an MRI evaluation in the future;
9. Patient is not willing to maintain current medication regimen;
10. Female candidates of child bearing potential who are pregnant (confirmed by positive urine/blood pregnancy test), not using adequate contraception as determined by the investigator, or nursing (lactating) a child.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | End of 6 week stimulation trial
  The Fibromyalgia Impact Questionnaire (FIQ) is a self administered scale that was developed to measure fibromyalgia patient status, progress and outcomes. It measures the components of health that are most affected by fibromyalgia. The maximum score is 100 and a higher score indicates a greater impact of the syndrome on the person.
  The change in the Fibromyalgia Impact Questionnaire (FIQ) will be analyzed and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Diaz, Study Director — Abbott Medical Devices
Locations (1):
- Universitair Ziekenhuis Antwerpen, Antwerp, Belgium